CLINICAL TRIAL: NCT07032532
Title: An Open-Label, Single-Arm, Phase 2 Study to Evaluate the Efficacy and Safety of Golidocitinib in First-Line Therapy of Peripheral T-Cell Lymphoma
Brief Title: Assessing An Oral JAK1 Inhibitor, Golidocitinib, in Patients Who Have Newly Diagnosed Peripheral T-Cell Lymphoma (JACKPOT23)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huiqiang Huang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2024J0002
Record Dates: First submitted 2025-05-19; First posted 2025-06-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Golidocitinib monotherapy or Golidocitinib in combination with CHOP (Experimental): During induction therapy, eligible patients will receive golidocitinib 150mg orally once daily for 6 induction cycles and then undergo restaging (PET/CT scan). Patients that achieve CR will continue golidocitinib monotherapy for 6 more cycles at the previously described dose; patients that achieve PR or SD will receive golidocitinib 150 mg every other day in combination with CHOP for 6 cycles. The maintenance therapy starts at Cycle 13 Day 1 and will consist of golidocitinib at 150 mg once daily for up to 1 year in patients that achieve CR, or continue until disease progression, unacceptable toxicity, death, withdrawal of consent, or the study is terminated by the investigator and/or IND sponsor for PR/SD patients . A treatment cycle consists of 21 days.
  Interventions: Drug: Golidocitinib; Drug: Golidocitinib plus CHOP

INTERVENTIONS:
Drug: Golidocitinib — Golidocitinib 150mg orally once daily in a 21-day cycle
Drug: Golidocitinib plus CHOP — Golidocitinib 150mg orally every other day with CHOP (Cyclophosphamide: 750mg/m2, IV, d1 ; Doxorubicin: 50mg/m2, IV, d1; Vincristine: 1.4mg/m2, IV, d1 ; Prednison: 100mg, po, d1-5) in a 21-day cycle for 6 cycles.

SUMMARY:
This study will treat patients with newly diagnosed PTCL, who have no prior systemic treatment for T-cell lymphoma. This study will assess the anti-tumor efficacy of golidocitinib using 2-year Progression-Free Survival rate as primary endpoint. In addition, it will help to understand what type of side effects may occur with the drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18 years old.
2. ECOG performance status 0-2 with no deterioration over the previous 2 weeks.
3. Predicted life expectancy ≥ 12 weeks.
4. Patients must have histologically confirmed peripheral T-cell lymphoma. Eligible histological subtypes are restricted to the following:

   * PTCL, not otherwise specified (PTCL, NOS) (the proportion of PTCL-NOS subtype will not exceed 30% of all enrolled)
   * Angioimmunoblastic T-cell lymphoma (AITL)
   * Follicular T cell lymphoma
   * PTCL with T follicular helper (TFH) phenotype
5. Patients must have measurable disease according to the 2014 Lugano classification.
6. Patients must be treatment naïve with no prior systemic treatment for T-cell lymphoma.
7. Adequate bone marrow reserve and organ system functions.
8. Willing to comply with contraceptive restrictions.

Exclusion Criteria:

1. Intervention with any of the following:

   * Any investigational anti-cancer agents or study anti-cancer drugs from a previous clinical study.
   * Any cytotoxic chemotherapy from a previous treatment regimen.
   * Corticosteroids at dosages equivalent to prednisone > 40 mg/day within 7 days.
2. Major surgery procedure, or significant traumatic injury within 4 weeks.
3. Prior treatment with a JAK or STAT3 inhibitor.
4. Prior treatment with any onco-immunotherapy in 28 days.
5. Live vaccines within 28 days.
6. Patients currently receiving (or unable to stop use at least 14 days prior to receiving the first dose) medications or herbal supplements known to be Potent inhibitors or inducers of CYP3A.
7. Central nervous system or leptomeningeal lymphoma.
8. Past medical history of pneumonitis, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
9. Patients with disease condition which requires the treatment of immunosuppressants, biologics, or NSAID.
10. Active infections
11. Clinically significant cardiac disorders or abnormalities. Acute thrombotic diseases within 90 days.
12. Another malignancy within 5 years prior to enrollment with the exception of adequately treated in-situ carcinoma of the cervix, uterus, basal or squamous cell carcinoma or nonmelanomatous skin cancer.
13. Gastrointestinal disorders that is inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of golidocitinib.
14. History of hypersensitivity to active or inactive excipients of golidocitinib or drugs with a similar chemical structure or class.
15. Women who are breast feeding or pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
2-year Progression-Free Survival Rate | Approximately 3.5 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 3.5 years
Complete Response Rate (CRR) | Approximately 3.5 years
Duration of response (DoR) | Approximately 3.5 years
Progression-Free Survival (PFS) | Approximately 3.5 years
Time To Response (TTR) | Approximately 3.5 years
Overall Survival (OS) | Approximately 3.5 years

OTHER OUTCOMES:
Incidence of adverse events | Approximately 3.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No